CLINICAL TRIAL: NCT00306852
Title: Tube Versus Trabeculectomy (TVT) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Pfizer (Industry); Abbott Medical Optics (Industry)
Responsible Party: Principal Investigator, Steven J. Gedde, Professor of Ophthalmology, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19990167
Record Dates: First submitted 2006-03-23; First posted 2006-03-24 (Estimated); Results first posted 2015-11-25 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-10

CONDITIONS: Glaucoma
Keywords: Glaucoma; Trabeculectomy; Tube shunt surgery
MeSH Terms: conditions — Glaucoma | interventions — Glaucoma Drainage Implants; Trabeculectomy; Mitomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trabeculectomy (Active Comparator): Trabeculectomy with mitomycin C
  Interventions: Procedure: Trabeculectomy with mitomycin C
- Implant (Active Comparator): Baerveldt Implant
  Interventions: Procedure: Baerveldt implant

INTERVENTIONS:
Procedure: Baerveldt implant — Patients will be randomized to receive a 350 mm^2 Baerveldt glaucoma implant or a Trabeculectomy (guarded filtration surgery) with mitomycin C (0.4 mg/ml for 4 minutes)
  Arms: Implant
Procedure: Trabeculectomy with mitomycin C — Patients will be randomized to receive either a Trabeculectomy (guarded filtration surgery) with mitomycin C (0.4 mg/ml for 4 minutes) or a 350 mm^2 Baerveldt glaucoma implant
  Arms: Trabeculectomy

SUMMARY:
The purpose of the Tube Versus Trabeculectomy (TVT) Study is to compare the safety and efficacy of nonvalved tube shunt surgery to trabeculectomy with mitomycin C in patients with previous ocular surgery.

DETAILED DESCRIPTION:
Glaucoma surgery is performed when further intraocular pressure (IOP) reduction is needed despite the use of maximum tolerated medical therapy and appropriate laser treatment. Trabeculectomy is generally used as the initial incisional surgical procedure in managing glaucoma. However, eyes in which trabeculectomy has failed are at greater risk of failure with subsequent filtering surgery. Wound modulation with antifibrotic agents, like mitomycin C (MMC) and 5-fluorouracil (5-FU), has been shown to increase the success rate of trabeculectomy in eyes that have undergone previous ocular surgery. Although antifibrotic agents have increased the likelihood of IOP control following filtering surgery, they have also increased the risk of complications. The prevalence of bleb leaks, bleb-related infections, and bleb dysesthesia associated with a perilimbal filtering bleb suggests the need to consider alternatives. Tube shunts (or glaucoma drainage implants) offer an alternative to trabeculectomy in the surgical management of glaucoma, and these devices have been growing in popularity in recent years.

Practice patterns vary in the surgical management of glaucoma in eyes with previous ocular surgery. In 1996, Chen and colleagues conducted an anonymous survey of members of the American Glaucoma Society (AGS) and Japanese Glaucoma Society (JGS) to evaluate use of antifibrotic agents and tube shunts. The survey presented ten clinical situations requiring glaucoma surgical intervention. The majority of respondents (59-83%) preferred trabeculectomy with MMC for the clinical scenarios involving prior ocular surgery, although many of those surveyed elected to use a tube shunt, trabeculectomy with 5-FU, or trabeculectomy without an antifibrotic agent. In 2002, Joshi and associates re-administered the same survey to members of the AGS. Respondents still favored trabeculectomy with MMC, but the percentage usage of tube shunts had significantly increased. The greatest practice pattern shift was observed in patients with previous cataract and glaucoma surgery. In particular, selection of tube shunts as the preferred surgical approach increased from 7% to 22% in eyes with prior trabeculectomy, and increased from 8% to 22% in eyes with prior extracapsular or intracapsular cataract extraction.

The lack of consensus among glaucoma surgeons regarding the use of tube shunts or trabeculectomy with an antifibrotic agent in eyes that have had prior cataract or glaucoma surgery likely relates to the fact that available clinical data has not shown one surgical procedure to be superior to the other. Similar surgical results have been reported with both glaucoma procedures in eyes with aphakia/pseudophakia and failed filters when studied separately. Success rates have ranged from 50% to 88% for tube shunts, and 48% to 86% for filtering surgery with an antifibrotic agent in case series studying aphakic/pseudophakic eyes. Success rates have ranged from 44% to 88% for tube shunts, and 61% to 100% for 5-FU and MMC trabeculectomy in eyes with failed filters. Comparable rates of severe complications have also been reported with tube shunt surgery and trabeculectomy with an adjunctive antifibrotic agent.

The Tube Versus Trabeculectomy (TVT) Study was designed to prospectively compare the safety and efficacy of nonvalved tube shunt surgery and trabeculectomy with MMC. Patients with uncontrolled glaucoma who had prior cataract extraction with intraocular lens implantation and/or failed filtering surgery were enrolled in this multicenter clinical trial and randomized to placement of a 350 Baerveldt glaucoma implant (Advanced Medical Optics, Irvine, CA) or trabeculectomy with MMC (0.4 mg/ml for 4 minutes). The goal of this investigator initiated trial is to provide information that will assist in surgical decision-making in similar patient groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85 years
* Intraocular pressure greater than or equal to 18 mm Hg and less than or equal to 40 mm Hg
* Previous trabeculectomy, cataract extraction with intraocular lens implantation, or both

Exclusion Criteria:

* Unwilling or unable to give consent, unwilling to accept randomization, or unable to return for scheduled protocol visits
* Pregnant or nursing women
* No light perception vision
* Active iris neovascularization or active proliferative retinopathy
* Iridocorneal endothelial syndrome
* Epithelial or fibrous downgrowth
* Aphakia
* Vitreous in the anterior chamber for which a vitrectomy is anticipated
* Chronic or recurrent uveitis
* Severe posterior blepharitis
* Unwilling to discontinue contact lens use after surgery
* Previous cyclodestructive procedure, scleral buckling procedure, or presence of silicone oil
* Conjunctival scarring precluding a trabeculectomy superiorly
* Need for glaucoma surgery combined with other ocular procedures (eg cataract surgery, penetrating keratoplasty, or retinal surgery) or anticipated need for additional ocular surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 1999-10; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Gedde, M.D., Study Chair — Bascom Palmer Eye Institute; Dale K Heuer, M.D., Study Chair — Medical College of Wisconsin; Richard K Parrish, M.D., Study Chair — Bascom Palmer Eye Institute
Locations (17):
- United States (16):
  - Scripps Clinic, La Jolla, California
  - University of Southern California, Los Angeles, California
  - University of California Davis, Sacramento, California
  - University of Florida, Gainesville, Florida
  - Bascom Palmer Eye Institute, Miami, Florida
  - Loyola University, Maywood, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Louis University, St Louis, Missouri
  - New York Eye and Ear Infirmary, New York, New York
  - Duke University, Durham, North Carolina
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas Houston, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Moorfields Eye Hospital, London, United Kingdom

REFERENCES:
- [Derived] Vanner EA, Sun CQ, McSoley MJ, Persad PJ, Feuer WJ, Lum F, Kelly SP, Parrish RK, Chang TC, Gedde SJ. Tube Versus Trabeculectomy IRISⓇ Registry 1-Year Composite Outcome Analysis with Comparisons to the Randomized Controlled Trial. Am J Ophthalmol. 2021 Jul;227:87-99. doi: 10.1016/j.ajo.2021.02.023. Epub 2021 Feb 28. PMID 33657420
- [Derived] Saheb H, Gedde SJ, Schiffman JC, Feuer WJ; Tube Versus Trabeculectomy Study Group. Outcomes of glaucoma reoperations in the Tube Versus Trabeculectomy (TVT) Study. Am J Ophthalmol. 2014 Jun;157(6):1179-1189.e2. doi: 10.1016/j.ajo.2014.02.027. Epub 2014 Feb 14. PMID 24531027
- [Derived] Gedde SJ, Schiffman JC, Feuer WJ, Herndon LW, Brandt JD, Budenz DL; Tube versus Trabeculectomy Study Group. Treatment outcomes in the Tube Versus Trabeculectomy (TVT) study after five years of follow-up. Am J Ophthalmol. 2012 May;153(5):789-803.e2. doi: 10.1016/j.ajo.2011.10.026. Epub 2012 Jan 15. PMID 22245458
- [Derived] Gedde SJ, Herndon LW, Brandt JD, Budenz DL, Feuer WJ, Schiffman JC; Tube Versus Trabeculectomy Study Group. Postoperative complications in the Tube Versus Trabeculectomy (TVT) study during five years of follow-up. Am J Ophthalmol. 2012 May;153(5):804-814.e1. doi: 10.1016/j.ajo.2011.10.024. Epub 2012 Jan 14. PMID 22244522
- [Derived] Gedde SJ, Schiffman JC, Feuer WJ, Herndon LW, Brandt JD, Budenz DL; Tube Versus Trabeculectomy Study Group. Three-year follow-up of the tube versus trabeculectomy study. Am J Ophthalmol. 2009 Nov;148(5):670-84. doi: 10.1016/j.ajo.2009.06.018. Epub 2009 Aug 11. PMID 19674729

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Trabeculectomy | Implant
Started | 105 | 107
Completed | 76 | 69
Not Completed | 29 | 38
Not completed — Death | 14 | 14
Not completed — Lost to Follow-up | 15 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Trabeculectomy | Implant | Total
Number analyzed (Participants) | 105 | 107 | 212
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (9.9) | 70.9 (11.0) | 71.0 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 64 | 112
  Male | 57 | 43 | 100
Intra-ocular pressure (IOP) [Mean (Standard Deviation); unit: mm Hg] | 25.6 (503) | 25.1 (5.3) | 25.3 (5.3)
GLAUCOMA MEDICATIONS [Mean (Standard Deviation); unit: number of medications used] | 3.0 (1.2) | 3.2 (1.1) | 3.1 (1.2)
ETDRS (Early Treatment Diabetic Retinopathy Study) VISUAL ACUITY [Mean (Standard Deviation); unit: Letters] — Numbers of letters read correctly on the ETDRS (Early Treatment Diabetic Retinopathy Study) chart.
  Letters | 64.4 (19.6) | 62.7 (24.1) | 63.6 (21.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Intraocular Pressure
Description: The data value from the Baseline visit and 5 year follow-up visit were combined. Specifically, values were calculated by subtracting the 5 Year Intraocular Pressure from the Baseline Intraocular Pressure.
Time Frame: Baseline to 5 years
Population: Participants who completed 5 years of follow-up
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Trabeculectomy | Implant
Number analyzed (Participants) | 63 | 61
mm Hg | 12.6 (5.9) | 14.4 (6.9)

2. Primary Outcome: Rate of Complications
Description: Complications associated with both surgical procedures
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Trabeculectomy | Implant
Number analyzed (Participants) | 105 | 105
participants
  EARLY POSTOPERATIVE COMPLICATIONS | 39 | 33
  LATE POSTOPERATIVE COMPLICATIONS | 38 | 36

3. Secondary Outcome: Visual Acuity
Description: Visual acuity was measured by the total number of letters read (correctly) using a ETDRS eye chart
Time Frame: 5 years
Population: Participants who complete 5 years of follow-up
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Trabeculectomy | Implant
Number analyzed (Participants) | 41 | 37
Letters
  PATIENTS WITH COMPLICATIONS | 56 (26) | 33 (31)
  PATIENTS WITHOUT COMPLICATIONS | 44 (30) | 46 (36)

4. Secondary Outcome: Reoperations for Glaucoma
Description: Reoperations for glaucoma was defined as additional glaucoma surgery requiring a return to the operating room.
Time Frame: 5 years
Measure: Number; unit: participants
Arm/Group | Trabeculectomy | Implant
Number analyzed (Participants) | 105 | 107
participants | 15 | 20

5. Secondary Outcome: Need for Supplemental Medical Therapy
Description: The number of supplemental glaucoma medications required in the Implant Group and Trabeculectomy Group at 5 years
Time Frame: 5 years
Measure: Mean (Standard Deviation); unit: number of medications
Arm/Group | Trabeculectomy | Implant
Number analyzed (Participants) | 105 | 107
number of medications | 1.2 (1.5) | 1.4 (1.3)

6. Secondary Outcome: Failure Rate
Description: Failure was prospectively defined as IOP greater than 21 mm Hg or less than 20 percent reduction below baseline on 2 consecutive follow-up visits after 3 months, IOP less than or equal to 5 mm Hg on 2 consecutive follow-up visits after 3 months, re-operation for glaucoma, or loss of light perception vision.
Time Frame: 5 years
Measure: Number; unit: percentage of participants
Arm/Group | Trabeculectomy | Implant
Number analyzed (Participants) | 105 | 107
percentage of participants | 46.9 | 29.8

ADVERSE EVENTS:
Arm/Group | Trabeculectomy | Implant
Serious Adverse Events (participants affected / at risk) | 13/105 | 15/107
Other Adverse Events (participants affected / at risk) | 77/105 | 58/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Trabeculectomy (N=105) | Implant (N=107)
CANCER (General disorders) | 2 | 0 — Specific Cancer type or cause - unknown.
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
STROKE (Vascular disorders) | 1 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 0 | 1
UNKNOWN CAUSE OF DEATH (General disorders) | 7 | 6 — Study Team/Coordinating Center was unable to obtain the specific cause of death for 12 Subjects.
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1
LUNG CANCER (Respiratory, thoracic and mediastinal disorders) | 1 | 0
BONE CANCER (Musculoskeletal and connective tissue disorders) | 0 | 1 — CLASSIFICATION UNKNOWN
MYCARDIAL INFRACTION (Cardiac disorders) | 0 | 4
CORONARY ARTERY BYPASS SURGERY (Surgical and medical procedures) | 0 | 1 — MORE SPECIFIC CAUSE OF DEATH UNAVAILABLE.
SQUAMOUS CELL CARCINOMA OF THE TRACHEA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Trabeculectomy (N=105) | Implant (N=107)
CHOROIDAL EFFUSION (Eye disorders) | 18 | 17
SHALLOW OR FLAT ANTERIOR CHAMBER (Eye disorders) | 10 | 12
WOUND LEAK (Eye disorders) | 12 | 1
HYPHEMA (Eye disorders) | 8 | 2
AQUEOUS MISDIRECTION (Eye disorders) | 1 | 3
SUPRACHOROIDAL HEMORRHAGE (Eye disorders) | 3 | 2
VITREOUS HEMORRHAGE (Eye disorders) | 1 | 1
DECOMPRESSION RETINOPATHY (Eye disorders) | 1 | 0
CYSTOID MACULAR EDEMA (Eye disorders) | 3 | 5
PERSISTENT CORNEAL EDEMA (Eye disorders) | 9 | 17
DYSESTHESIA (Eye disorders) | 8 | 1
PERSISTENT DIPLOPIA (Eye disorders) | 2 | 6
ENCAPSULATED BLEB (Eye disorders) | 6 | 2
BLEB LEAK (Eye disorders) | 6 | 0
HYPOTONY MACULOPATHY (Eye disorders) | 5 | 1
TUBE EROSION (Eye disorders) | 0/0 | 5
ENDOPHTHALMITIS/BLEBITIS (Eye disorders) | 5 | 1
CHRONIC OR RECURRENT IRITIS (Eye disorders) | 1 | 2
TUBE OBSTRUCTION (Eye disorders) | 0/0 | 6
RETINAL DETACHMENT (Eye disorders) | 1 | 1
CORNEAL ULCER (Eye disorders) | 1 | 0
SERIOUS COMPLICATIONS (Eye disorders) | 21 | 24 — Serious complications were defined as postoperative complications requiring a re-operation to manage the complication and/or resulting in loss of 2 or more lines of Snellen VA.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No